CLINICAL TRIAL: NCT06829394
Title: A Type 1 Hybrid Effectiveness-Implementation Evaluation of a City-Level Transitional Housing Program's Effects on Health, Economic, and Psychologic Outcomes Among People With HIV
Brief Title: Transitional Housing and HIV Health
Status: Recruiting | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: Philadelphia Department of Public Health (Other Government)
Responsible Party: Sponsor
Other Study IDs: 855009
Record Dates: First submitted 2025-01-28; First posted 2025-02-17 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: HIV; HIV Antiretroviral Therapy (ART) Adherence; Housing Instability
Keywords: HIV; Housing; Structural Interventions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Arms Around You Program Waitlist: These are individuals that are part of the lottery but not yet assigned to the program.
- Arms Around You Program Recipients: These are individuals that were part of the lottery AND assigned to the program
  Interventions: Other: Program Assignment

INTERVENTIONS:
Other: Program Assignment — The intervention group will include People living with HIV who were assigned to the Arms Around You Program in the lottery.
  Groups: Arms Around You Program Recipients

SUMMARY:
The goal of this pilot study is to evaluate the implementation and outcomes of the Arms Around You (AAY) program, a supportive housing initiative launched by the Philadelphia Department of Public Health (PDPH) in 2024. The program aims to address housing instability among people with HIV (PWH) using a Housing First model. The main questions it seeks to answer are:

1. How does AAY affect HIV-related outcomes, particularly viral suppression and antiretroviral therapy (ART) adherence?
2. What are the program's effects on economic, psychological, and secondary health outcomes?
3. How feasible, acceptable, and scalable is the program for broader implementation? Participants will be assigned to immediate program access or a waitlist using a random lottery system, creating treatment and control groups, respectively. Surveys and health data will be collected at baseline and over 36 months to assess changes in outcomes such as viral suppression, housing security, mental health, and financial well-being. Qualitative interviews with participants and stakeholders will complement quantitative findings to explore mechanisms of change and guide program optimization.

DETAILED DESCRIPTION:
Housing instability significantly impedes HIV-related outcomes, such as engagement in care, ART adherence, and viral suppression. Structural racism and poverty exacerbate these disparities, particularly for racial and sexual minorities. To address this, the PDPH developed the AAY program, which combines rent support (up to 48 months), housing medical case management (MCM), and intensive housing counseling, following client-centered, harm-reduction principles.

This hybrid type 1 effectiveness-implementation study will evaluate the effects of the AAY intervention on health, economic, and psychological outcomes. PWH experiencing homelessness or severe housing instability will be prioritized for the program. The lottery-based design will allow researchers to observe differences between those granted immediate program access and those on the waitlist (who will receive standard of care treatment and serve as the control group). The primary outcomes of interest are HIV viral suppression (defined as <200 copies/mL) and ART adherence, measured via pharmacy refill data. Secondary outcomes include housing security, food security, financial stress, psychological distress, and health-related quality of life.

Researchers will use mixed methods to collect data over 36 months. Quantitative data will include pre- and post-program surveys, pharmacy refill records, and PDPH surveillance data. Qualitative data will be gathered through semi-structured interviews with key stakeholders, including program participants, waitlisted individuals, housing MCMs, and city leaders. These interviews will explore the program's acceptability, implementation challenges, and pathways through which housing support influences HIV outcomes.

Approximately 200 participants will be enrolled in the survey study, with data collected at baseline and at 6, 12, 24, and 36 months. Key implementation outcomes, such as the program's reach, sustainment, and costs, will also be analyzed to inform scalability. This study will provide critical evidence on how housing interventions can reduce health inequities and improve HIV-related outcomes, offering actionable insights for policymakers and public health leaders in Philadelphia and beyond.

ELIGIBILITY:
Inclusion Criteria: Inclusion criteria for the Lottery Population will be all PWH in priority group 2 included in the initial lottery for access to the AAY program.

Inclusion criteria for the Survey population is (1) eligible for the HIV transitional housing program (2) priority group 2 with anticipated inclusion in the inital lottery (3) no plans to leave Philadelphia in the next year (4) regular access to a telephone to be able to complete phone surveys (5) able to provide informed consent.

-

Exclusion Criteria: Does not meet the above inclusion criteria.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People living with HIV in Priority Group 2 (at high risk for eviction/homelessness) who participate in the lottery, and a smaller sub-population of PWH who participate in the study surveys.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-02-25 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
HIV viral suppression - defined as HIV RNA < 200 copies/mL | From lottery to 12 months after the lottery
  HIV viral suppression during two discrete 6-month periods after the lottery for access to the AAY program. (Lottery population)
ART adherence | During discrete 3-month periods up to 12 months after the lottery
  ART adherence (survey population)

SECONDARY OUTCOMES:
Engagement in HIV care | From lottery to 12 months after the lottery
  Engagement in HIV care (defined as having an HIV viral load or CD4 count measured within a 6-month period). (Lottery Population)
Health Related Quality of Life | 6, 12, 24 and 36 months after assignment to the lottery
  CDC HRQOL-4 (Survey Population). A 4-question scale that assesses four key domains: self-rated general health, physical health, mental health, and activity limitations. Higher score is better outcome.
Alcohol use | 6, 12, 24 and 36 months after assignment to the lottery
  Alcohol Use Disorders Identification Test-Concise: AUDIT-C (Survey Population). Scored on a scale 0-12 with a higher score indicative of a worse outcome.
Cigarette Dependence | 6, 12, 24 and 36 months after assignment to the lottery
  Cigarette Dependence Scale: CDS-5 (Survey Population). Scored on a scale 1-5
Recent Substance Use | 6, 12, 24 and 36 months after assignment to the lottery
  National Institute on Drug Abuse. Screening for Drug Abuse in General Medical Settings. (Survey Population)
ED visits and reason for most recent visit | 6, 12, 24 and 36 months after assignment to the lottery
  (Survey Population)
Hospitalizations | 6, 12, 24 and 36 months after assignment to the lottery
  (Survey Population)
Out of pocket health costs | 6, 12, 24 and 36 months after assignment to the lottery
  Outpatient, ED/inpatient, prescription, other (survey population)
HIV Transmission risk behaviors | 6, 12, 24 and 36 months after assignment to the lottery
  (survey population)
Housing security | 6, 12, 24 and 36 months after assignment to the lottery
  US Census Bureau. 2019 American Housing Survey Instrument Items. (Survey population)
Perceived Housing Quality | 6, 12, 24 and 36 months after assignment to the lottery
  Cerin E, Saelens BE, Sallis JF, Frank LD. Neighborhood Environment Walkability Scale (survey population)
Neighborhood safety scale | 6, 12, 24 and 36 months after assignment to the lottery
  Housing Satisfaction for Persons with Psychiatric Disabilities (survey population)
Income as % federal poverty level | 6, 12, 24 and 36 months after assignment to the lottery
  (survey population)
Current employment status | 6, 12, 24 and 36 months after assignment to the lottery
  (survey population)
Participation in other public programs (e.g. SNAP, Medicaid) | 6, 12, 24 and 36 months after assignment to the lottery
  (survey population)
Financial Stress | 6, 12, 24 and 36 months after assignment to the lottery
  CFPB (survey population)
Food Security | 6, 12, 24 and 36 months after assignment to the lottery
  USDA (survey population)
Stress | 6, 12, 24 and 36 months after assignment to the lottery
  Perceived Stress Scale (survey population)
Psychological Distress | 6, 12, 24 and 36 months after assignment to the lottery
  Kessler 6+ (survey population)
Hope | 6, 12, 24 and 36 months after assignment to the lottery
  State Hope Scale (Survey population). 8-item scale
Preferences survey | 6, 12, 24 and 36 months after assignment to the lottery
  Preference Survey Probabilistic Scale (survey population). Scale 0-10 with higher number indicating better outcome.
Time preference: Hyperbolicity | 6, 12, 24 and 36 months after assignment to the lottery
  Brownback incentivized questions (survey population)
Time Preferences: Patience | 6, 12, 24 and 36 months after assignment to the lottery
  Brownback incentivized questions (survey population)
Time Horizon | 6, 12, 24 and 36 months after assignment to the lottery
  Laajaj (survey population)
HIV Stigma | 6, 12, 24 and 36 months after assignment to the lottery
  HIV stigma scale, short form (survey population)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No